CLINICAL TRIAL: NCT01377441
Title: Randomized, Double-blind, Pilot Study on the Effect of Intravenous Ibuprofen on Inflammatory Responses in Patients Undergoing Surgery With General Anesthesia: Correlation With Clinical Outcomes
Brief Title: Effect of Intravenous Ibuprofen on Inflammatory Responses in Patients Undergoing Surgery With General Anesthesia.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Samples lost during Hurricane Sandy. Study now taking place at other medical centers.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-01188
Record Dates: First submitted 2011-06-17; First posted 2011-06-21 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-11

CONDITIONS: Inflammatory Response
Keywords: Ibuprofen; Cytokines; Recovery; IV ibuprofen; major surgery
MeSH Terms: interventions — Ibuprofen; Anti-Inflammatory Agents, Non-Steroidal; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ibuprofen (Experimental): Eligible subjects will be randomized to one of the two treatment group in a 1:1 ratio to receive either IV ibuprofen or matching placebo.
  Interventions: Drug: Ibuprofen
- Placebo/Saline solution (Placebo Comparator): Eligible subjects will be randomized to one of the two treatment group in a 1:1 ratio to receive either IV ibuprofen or matching placebo
  Interventions: Drug: Placebo/Saline solution

INTERVENTIONS:
Drug: Ibuprofen — Patients will receive either 800mg IV ibuprofen or placebo pre-operatively. Post-operatively, patients will receive either 800mg IV ibuprofen or placebo 6 hours after the first dose.
  Other Names: nonsteroidal anti-inflammatory drug (NSAID)
  Arms: Ibuprofen
Drug: Placebo/Saline solution — Patients will receive placebo pre-operatively. Post-operatively, patients will receive placebo at least 6 hours after the initial dose.
  Arms: Placebo/Saline solution

SUMMARY:
The administration of anti-inflammatory drugs such as ibuprofen before and after surgery has not been studied extensively. Subjects are being asked to participate in this study because they are scheduled for surgery and because the investigators want to study ways to improve recovery from surgery. Ibuprofen will be given several times before and after surgery. The investigators will ask questions to determine recovery and the investigators will draw blood to determine inflammatory response.

DETAILED DESCRIPTION:
Human and animal studies suggest cyclooxygenase-inhibitors (COX-inhibitors) decrease the production of inflammatory mediators. Studies also suggest that COX inhibitors attenuate increases in corticosterone and eicosanoid levels after endotoxin injection. COX inhibitors also appear to have anticancer effects, inhibiting angiogenesis, tumor growth, and metastatic burden. These results suggest a role for IV ibuprofen in preventing untoward inflammatory responses, shortening post-surgical convalescence, improving patient satisfaction, and reducing the rate of complications occurring during the recovery from surgery. However, there are no studies that have evaluated the relationship between administration of IV ibuprofen, ensuing immunomodulation, and long-term outcomes.

Study Objective. The aim of the proposed study is to examine the effect of intravenous(IV) ibuprofen on the inflammatory response in major surgery. More importantly, the investigators will correlate changes in the concentration of inflammatory mediators with meaningful clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, 18 and over, who will undergo surgery lasting longer than one hour with general anesthesia
2. Subject is non-lactating and is either:

   * Not of childbearing potential
   * Of childbearing potential but is not pregnant at time of baseline as determined by pre-surgical pregnancy testing.
3. Subject is ASA physical status 1, 2, or 3

Exclusion Criteria:

1. Cognitively impaired (by history)
2. Subject requires chronic antipsychotic history
3. Subject is anticipated to require an additional surgery within 90 days after the intended surgery
4. Chronic use of steroids or opioids
5. Subject has received treatment with COX inhibitors within 3 days of study entry
6. Subject for whom opiates, benzodiazepines, and COX inhibitors are contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Doan, MD, Principal Investigator — NYU Langone Medical Center
Locations (2):
- United States (2):
  - NY Methodist Hospital, Brooklyn, New York
  - NYU Langone Medical Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the perioperative area.
Groups:
- Ibuprofen: Eligible subjects will be randomized to one of the two treatment group in a 1:1 ratio to receive either IV ibuprofen or matching placebo.
  Ibuprofen: Patients will receive either 800mg IV ibuprofen or placebo pre-operatively.
  Post-operatively, patients will receive either 800mg IV ibuprofen or placebo 6 hours after the first dose.
Period: Overall Study
Arm/Group | Ibuprofen | Placebo/Saline Solution
Started | 0 | 0
Completed | 0 (All data for this study was lost after Hurricane Sandy.) | 0 (All data for this study was lost after Hurricane Sandy.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All data was lost after Hurricane Sandy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibuprofen | Placebo/Saline Solution | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: Concentrations of the Cytokines Tumor Necrosis Factor Alpha (TNF-alpha), Interleukin IL-1Beta (IL-1Beta), IL-2, IL-6, IL-10, and Interferon-gamma (IFN-gamma) as Well as Prostaglandin E2 at Different Time Points.
Description: Concentration of the cytokines TNF-alpha, IL-1Beta, IL-2, IL-6, IL-10, and IFN-gamma as well as prostaglandin E2 at different time points will be our primary outcome. Changes in mediator levels in the IV ibuprofen versus placebo groups will be compared. Plasma samples will be collected before administration of any drug (after placement of IV lines), at the end of the surgery, and on the first postoperative day.
Time Frame: 48h
Population: Unfortunately, due to major flooding at our site, due to Hurricane Sandy, all data and samples for this study were lost. Therefore, it was impossible to analyze any data for this study.
Arm/Group | Ibuprofen | Placebo/Saline Solution
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Quality of Recovery Score (QoR-40).
Description: The secondary outcome parameters will be the quality of recovery score (QoR-40) to measure quality of recovery from surgery, a simple fatigue scale, digits forward and backward, and the global depression schedule. Forty questions in five dimensions will be scored by patients on a five-point Likert scale. Seven point fatigue scales (in- and out-patient) is often used to assess progress of recovery in head trauma patients. Metrics will be administered on at the baseline visit and or on the day of surgery and on postoperative days 1, 2, 4 and 6.
Time Frame: 48h
Population: No data displayed because Outcome Measure has zero total participants analyzed.
Arm/Group | Ibuprofen | Placebo/Saline Solution
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Unfortunately, due to major flooding of our site during Hurricane Sandy, all data and samples for this study were lost. Therefore, no AE data is available.
Arm/Group | Ibuprofen | Placebo/Saline Solution
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No